CLINICAL TRIAL: NCT05596331
Title: SIRCUS : Social Information pRocessing in Children:an ocUlo-pupillometric Tool for Standard Evaluation
Brief Title: Social Information Processing in Children: an ocUlo-pupillometric Tool for Standard Evaluation
Acronym: SIRCUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Collaborators: UMR 1253, iBrain, Université de Tours, Inserm, Tours, France. (Unknown); Laboratory of Fundamental and Applied Computer Science of Tours, EA6300 (Unknown); National Research Agency, France (Other); Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DR220031/SIRCUS; 2022-A00870-43 (Registry Identifier: IDRCB)
Record Dates: First submitted 2022-09-08; First posted 2022-10-27 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group of adult subjects without ASD (Autism Spectrum Disorders) (Other): Age between 18 and 50 years
  Interventions: Other: eye-tracker
- Group of children without ASD (Other): Age between 2 and 12 years
  Interventions: Other: eye-tracker
- Group of children with ASD (Other): Age between 2 and 12 years Conformity with the diagnostic criteria of ASD according to DSM-V, ICD-10 or ICD-11
  Interventions: Other: eye-tracker
- Group of children without NDD (NeuroDevelopmental Disorders) (Other): Age between 0 and 12 years
  Interventions: Other: eye-tracker
- Group of children with NDD, or whose diagnosis is in progress (Other): Conformity to the diagnostic criteria of NDD
  Interventions: Other: eye-tracker

INTERVENTIONS:
Other: eye-tracker — Eye-tracker recordings of eye movements, gaze direction and pupillary reactivity

SUMMARY:
The goal of this observational study is to identify behavioral and physiological markers of social alterations in Autism Spectrum Disorders compared to Typically Developping peers. This single-centre study plan to use eye tracking to evaluate social disorders in Autism Spectrum Disorders (ASD). The investigators will estimate oculometric and pupillometric indices as potential ASD biomarkers. The study will last 4 years and will be organized in two phases.

DETAILED DESCRIPTION:
In a first phase (expected to last 12-16 months), after an experimental validation in typical adults, relevant oculometric and pupillometric indices will be identified in a typical population of children and in a clinically diagnosed population of ASD children.

In a second phase of the protocol (expected to last 32-36 months), biomarkers identified in the first phase will be tested on a larger population including other neurodevelopmental disorders.

ELIGIBILITY:
Inclusion Criteria:

Phase 1

All groups have these 2 criteria in common:

Free, informed and signed consent of both parents Enrolment in the social security system

The other criteria per group are as follows:

Group of adult subjects without ASD : Age between 18 and 50 years Group of children without ASD

* Age between 2 and 12 years
* Group of children with ASD Age between 2 and 12 years Conformity with the diagnostic criteria of ASD according to DSM-V, ICD-10 or ICD-11

Phase 2

* Group of children without TND : Age between 0 and 12 years
* Group of children with TND, or whose diagnosis is in progress (via PCO referral) :

Age between 0 and 12 years Conformity to the diagnostic criteria of TND

Exclusion Criteria:

Phase 1:

All groups have the 2 common exclusion criteria Known uncorrected visual pathologies Known personal neurological pathologies

And they have these criteria per group:

* Group of adult subjects without ASD: Subject under guardianship or trusteeship Diagnosis of ASD Group of children without ASD : Diagnosis of ASD
* Group of children with ASD ICD-10 diagnosis of PDD (Rett syndrome and Hayler syndrome) Phase 2
* Group of children without ASD : Diagnosis of ASD (confirmed or ongoing)

Ages: 1 Day to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 460 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2026-01-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Oculometric measurements 1: Tracking time | through study completion, an average of 1 year (first phase) and of 2 years (second phase)
  Mean of tracking time (ms) during entire stimuli duration
Oculometric measurements 2: Fixation time on the screen | through study completion, an average of 1 year (first phase) and of 2 years (second phase)
  Mean of fixation time on the screen (ms) during entire stimuli duration
Oculometric measurements 3: Fixation time on the eye area during entire stimuli duration | through study completion, an average of 1 year (first phase) and of 2 years (second phase)
  Mean of fixation time on the eye area of face stimuli (ms) during entire stimuli duration
Oculometric measurements 4: Fixation time on the mouth area of face stimuli | through study completion, an average of 1 year (first phase) and of 2 years (second phase)
  Mean of fixation time on the mouth area of face stimuli (ms) during entire stimuli duration
Pupillometric measurements | through study completion, an average of 1 year (first phase) and of 2 years (second phase)
  Mean of pupil dilation variation(mm) in response to entire stimuli duration
Discriminative power | through study completion, an average of 1 year (first phase) and of 2 years (second phase)
  AUROC (Area Under the Receiver Operating Characteristics, in percent) analysis of combined oculometric and pupillometric measurements. Scale score : 0-100% (above 70% : good performance; above 80% : excellent performance; above 90% : outstanding performance)

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Aguillon-Hernandez, MCU, Principal Investigator — UMR 1253, iBrain, Université de Tours, Inserm, Tours, France.
Locations (1):
- Service de Pédopsychiatrie-CHU-TOURS, Tours, France

IPD SHARING:
Plan to Share IPD: No